CLINICAL TRIAL: NCT00296842
Title: Prevention of Posttraumatic Stress Symptoms and Behavioral Problems in Children and Adolescents After Road Traffic Accidents: a Randomized Controlled Trial
Brief Title: Prevention of Posttraumatic Stress Symptoms and Behavioral Problems in Children After Road Traffic Accidents: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PICARTA-1
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Injury
Keywords: posttraumatic stress disorder; children; injury; road traffic accident
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Early psychological intervention — Psychoeducation, trauma narrative, provision of coping skills

SUMMARY:
The purpose of this study is to study the effectiveness of an early psychological intervention 7-10 days after a road traffic accident on posttraumatic stress and behavior of children and adolescents

DETAILED DESCRIPTION:
Within a randomized controlled design the effects of a brief psychological intervention (child, parents) after a road traffic accident shall be examined in a sample of 100 children and adolescents. After a baseline assessment 7-10 days after the accident participants are randomly assigned to an intervention or a control group. Both are re-assessed at 2 and 6 months after the accident by means of standardized questionnaires assessing posttraumatic stress symptoms, depression, and behavior.

ELIGIBILITY:
Inclusion Criteria:

Age 7-16 y Command of German language Road traffic accident inpatient or outpatient treatment at the University Children's Hospital Zurich no pretraumatic developmental delay

Exclusion Criteria:

severe head injury No command of the German language Age below 7 y or above 16 y Other major systemic illness

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2004-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
CAPS-CA | 10 days, 2 months, 6 months after intervention
CBCL | 10 days, 2 months, 6 months after intervention
DIKJ | 10 days, 2 months, 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Landolt, PhD, Principal Investigator — University Children's Hospital
Locations (1):
- University Children's Hospital, Psychosomatic and Psychiatry, Zurich, Switzerland

REFERENCES:
- [Result] Zehnder D, Meuli M, Landolt MA. Effectiveness of a single-session early psychological intervention for children after road traffic accidents: a randomised controlled trial. Child Adolesc Psychiatry Ment Health. 2010 Feb 8;4:7. doi: 10.1186/1753-2000-4-7. PMID 20181120